CLINICAL TRIAL: NCT03169296
Title: Clinical and Genomic Registry of Myelodysplastic Syndrome (MDS) and Secondary Acute Myeloid Leukaemia (AML) in Asia
Brief Title: Clinical and Genomic Registry of MDS in Asia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: AMWG001
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic syndrome; Mutations; Next-generation sequencing
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myelodysplastic syndrome (MDS) is a group of clonal haematopoietic stem cell disorders characterized by ineffective haematopoiesis leading to cytopenia, with a significant risk of progression to acute myeloid leukaemia (AML). Progression to AML and resistance to hypomethylating agents (HMA) are important unmet clinical needs. The pathophysiology of MDS and its progression to AML involve cytogenetic, genetic and epigenetic aberrations, and hence better understanding of the molecular landscape of MDS has important clinical implications. Also, future treatment strategies for MDS may involve exploitation of genetic information in designing more effective therapy encompassing single agents or combinatorial approaches.

The proposed cohort study aims to establish a registry of clinical and genomic registry of MDS and secondary AML in Asian patients, which allows the establishment of the mutational profile of patients and prognostic model for survival, as well as exploration of treatment strategies and prediction for treatment response.

DETAILED DESCRIPTION:
Myelodysplastic syndrome (MDS) is a group of clonal haematopoietic stem cell disorders characterized by ineffective haematopoiesis leading to cytopenia, with a significant risk of progression to acute myeloid leukaemia (AML). Conventional prognostic scoring of MDS is based on the degree of cytopenia, the percentage of bone marrow blast infiltration and karyotypic abnormalities. Risk categories based on prognostic scoring determine the therapeutic approaches. Treatment of high-risk MDS involves the use of hypomethylating agents (HMA), and allogeneic haematopoietic stem cell transplantation (HSCT) in younger patients. Clinical studies with HMAs including azacitidine and decitabine have shown a response rate of about 40% in high-risk patients, and median duration of response of merely 9 to 15 months. HMA failure is associated with a dismal outcome and a median survival of less than 5 months. Therefore, progression to AML and resistance to HMA are important unmet clinical needs.

The pathophysiology of MDS and its progression to AML involve cytogenetic, genetic and epigenetic aberrations. Genome-wide and targeted analyses from next-generation sequencing have identified mutations that may have prognostic and therapeutic significance. Recurrent mutations in more than 45 genes are found in over 85% of cases. Theses mutations are found in genes involved in DNA methylation (DNMT3A, TET2, IDH1/2), post-translational chromatin modification (EZH2, ASXL1), transcription regulation (TP53, RUNX1, GATA2), the RNA spliceosome machinery (SF3B1, U2AF1, SRSF2, ZRSR2), cohesion complexes (STAG2), and signal transduction (JAK2, KRAS, CBL). Mutations in TP53, EZH2, ETV6, RUNX1, SRSF2 and ASXL1 portend inferior survivals. Specific mutations, such as internal tandem duplications of FLT3 (FLT3-ITD), have been observed during disease progression and are potential therapeutic targets. Data arising from whole-genome sequencing (WGS) have shown that the clonal evolution of MDS to AML is dynamic and complex. The selection of clones during transformation is shaped by acquisition of genetic alterations during clonal expansion, as well as exposure to genotoxic chemotherapy.

Better understanding of the molecular landscape of MDS has important clinical implications. Firstly, prognosticating MDS based on molecular aberrations will supplement current models in stratifying patients for treatment. Secondly, molecular markers may better predict response and resistance to treatment with HMAs. Thirdly, detection of targetable molecular markers during treatment resistance or leukaemic transformation may provide an opportunity for specific therapy, as exemplified by the use of FLT3 inhibitors in FLT3-ITD positive secondary AML. Hence, future treatment strategies for MDS may involve exploitation of genetic information in designing more effective therapy encompassing single agents or combinatorial approaches. There are important gaps in knowledge in the field of MDS. First, there is currently no well-established model integrating molecular with clinicopathologic features in prognostic stratification. There is lack of large registry clinicopathologic and molecular information in Asian patients with MDS. To-date, there is paucity of data focusing on the impact of molecular aberrations on prognosis and treatment response.

The proposed cohort study aims to establish a registry of clinical and genomic registry of MDS and secondary AML in Asian patients, which allows the establishment of the mutational profile of patients and prognostic model for survival, as well as exploration of treatment strategies and prediction for treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is an adult at the time of diagnosis of MDS. An adult is a person who has attained the legally defined age in accordance with local law.
2. Both biological parents and all four biological grandparents of the subject are the original people of the Far East, Southeast Asia, or the Indian subcontinent.
3. Subject was diagnosed with one of the following disorders according to the World Health Organization (WHO) classification criteria 2016:

   1. Myelodysplastic syndrome (MDS)
   2. Chronic myelomonocytic leukaemia (CMML)
   3. MDS/ Myeloproliferative neoplasm (MPN) with ring sideroblasts and thrombocytosis (MPN-RS-T)
   4. MDS/MPN unclassifiable
4. In prospective and partial prospective/retrospective case, subject has provided a signed written informed consent of this study. In retrospective case, subject has previously provided a signed written informed consent on:

   1. voluntary provision of his/her data, and
   2. voluntary provision of archived/remaining specimens for genetic analysis, and
   3. authorizing storage and usage of archived/remaining specimens for any further analysis

Exclusion Criteria:

1. Subject was diagnosed with acute myeloid leukaemia under the WHO classification criteria 2016
2. Subject was diagnosed with myeloproliferative neoplasms under the WHO classification criteria 2016

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of MDS recruited is stated in the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to progression to secondary AML | 60 months
Overall survival | 60 months
Progression-free survival | 60 months

SECONDARY OUTCOMES:
Time to first response to hypomethylating agent treatment | 60 months
Best overall response to hypomethylating agent treatment | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Harinder Singh Harry Gill, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine, the University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No